CLINICAL TRIAL: NCT03791437
Title: Optimization of Chest Tube Drainage Management to Shorten Postoperative Hospital Stay and Increase Satisfaction of Patients After Video-Assisted Thoracic Surgery
Brief Title: Optimization of Chest Tube Drainage Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGMH-IRB-201701495A3
Record Dates: First submitted 2018-12-13; First posted 2019-01-02 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2022-03

CONDITIONS: Lung Diseases; Age >18 Years-old; Patient Who Received Thoracoscope Surgery
Keywords: digital chest tube system, shorten hospital stay
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: digital chest drainage system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment groups (Experimental): Post chest operative use Digital chest drainage system until Patient's discharge day
  Interventions: Device: Digital chest drainage system
- Control groups (Active Comparator): Post chest operative use traditional drainage system until Patient's discharge day Not use Digital chest drainage system
  Interventions: Device: Not use Digital chest drainage system

INTERVENTIONS:
Device: Digital chest drainage system — patients who received Digital chest drainage system
  Arms: Experiment groups
Device: Not use Digital chest drainage system — patients who not received Digital chest drainage system( traditional drainage system)
  Arms: Control groups

SUMMARY:
Early recovery after surgery was new developing science in recent years. However , there was few reports in thoracic surgery field . Investigators try to using digital chest drainage management system into the field of postoperative care and to see whether it could help patients to recovery from surgery as soon as possible. According to investigators's clinical data collecting , investigators will establish a new postoperative care guideline for those patients who receive thoracic surgery

DETAILED DESCRIPTION:
Drainage of the space between the ribs and lungs has been practiced since the time of Hippocrates. Thus far, the function of chest tubes, specifically to drain fluid or air from the pleural space, has virtually remained unchanged for more than 3000 years. The use of chest drainage tubes after thoracic surgery is crucial to evacuate air leakage and/or pleural effusion; however, delayed tube removal may exacerbate pain, delay recovery of lung function and prolong hospitalization. Recently, Thopaz digitally monitored thoracic drainage system (Medela Healthcare, Baar, Switzerland)has been designed to provide objective measurements of air leakage and pleural pressure. With this system, air leakage and pleural pressure can be accurately measured in mL/min and mm H2O, respectively. The rate of air leakage can be seen on a display in real time. Digital surveillance for air leakage is reported to reduce interobserver disagreement in decision making in the management of patients with chest tubes, which might help caregiver a more solid evidence of strategies of postoperative chest drainage care.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to join the study after thoroughly explanations
* Patient who received thoracoscope surgery for lung lesion

Exclusion Criteria:

* Not willing to join the study after thoroughly explanations
* Patients who have not received thoracoscope surgery for lung lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Air leak graph of digital drainage system | Follow patient 's condition in OPD post surgery in two years
  Compare Digital chest drainage system with traditional drainage system

SECONDARY OUTCOMES:
Days of hospital stay after surgery | Follow patient 's condition in OPD post surgery in two years
  Compare Digital chest drainage system with traditional drainage system

OTHER OUTCOMES:
Fluid graph of digital drainage system | Follow patient 's condition in OPD post surgery in two years
  Compare Digital chest drainage system with traditional drainage system
Patient Daily Activity | Until patient discharge from our hospital
  Using Wearable Device for monitor patient's sleep quality and activity

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Feng Wu, MD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan